CLINICAL TRIAL: NCT06861075
Title: CARPEUS : Effect of Carvedilol on the Portosystemic Gradient as Measured by Endoscopic Ultrasound
Acronym: CARPEUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOI 2023 POINCLOUX; 2024-518302-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-19; First posted 2025-03-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis; Portal Hypertension Related to Cirrhosis
Keywords: Carvedilol.; Portal hypertension in cirrhosis.; EUS-PPG measurement.
MeSH Terms: conditions — Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): All patients will receive Carvedilol per os (dose escalation up to 12.5 mg per day).
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol per os, day 1:3.125 mg once, day 2 to day 8: 6.25 mg/day (3.125 mg twice a day), day 9 to day 90 (end of study visit): 12.5 mg/day (6.25 mg twice a day).
  After the end of the study, treatment with Carvedilol will be prescribed by a cardiologist and continued at the dose of 12.5 mg/day.
  The follow-up of the patient will be then done according to the standard practice.
  Other Names: CARVEDILOL ARROW ® 6,25 mg

SUMMARY:
The purpose of this study is to assess the efficacy after one month of treatment with Carvedilol (12.5 mg daily) in primary prophylaxis of digestive haemorrhage due to portal hypertension in cirrhosis, by endoscopic ultrasound-guided portal pressure gradient measurement.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period to determine eligibility for entry study.

- Inclusion visit (day 1) includes an oesogastroduodenal fibroscopy (OGDF) followed by an endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement, an electrocardiogram, a clinical examination, and a first intake of study treatment : Carvedilol 3.125 mg.

Carvedilol, day 2 to day 8: 6.25 mg/day (3.125 mg twice a day). - Visit 2 (day 6 +/- 2 days): clinical examination, record of potential adverse events, vital signs (arterial pressure, pulse rate), electrocardiogram if indicated, assessment of compliance with study treatment.

Carvedilol, day 9 to day 90 (end of study visit): 12.5 mg/day (6.25 mg twice a day).

- Visit 3 (day 13 +/- 2 days): clinical examination, record of potential adverse events, vital signs (arterial pressure, pulse rate), electrocardiogram if indicated, assessment of compliance with study treatment.

Carvedilol will be continued at the dose of 12.5 mg/day, on a long-term basis. - Visit 4 (day 30-45): OGDF followed by an EUS-PPG measurement, clinical examination, record of potential adverse events, vital signs (arterial pressure, pulse rate), electrocardiogram if indicated, assessment of compliance with study treatment.

Carvedilol will be continued at the dose of 12.5 mg/day.

- Visit 5 (day 90 +/- 7 jours), end of study visit: clinical examination, record of potential adverse events, vital signs (arterial pressure, pulse rate), electrocardiogram, assessment of compliance with study treatment.

Treatment with Carvedilol will be prescribed by a cardiologist and continued at the dose of 12.5 mg/day.

Follow-up of the patient according to standard practice. NB: an adaptation of the dose of Carvedilol may be considered according to tolerability, throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Suspected portal hypertension associated with cirrhosis (of any aetiology) as defined by:

  1. Baveno VII criteria :

     Liver stiffness ≥ 25 kPa Or Liver stiffness between 20 and 25 kPa and platelets < 150 G/L Or Liver stiffness between 15 and 20 kPa and platelets < 110 G/L Or Liver stiffness > 20 kPa and/or platelets < 150 G/L in patients with cirrhosis due to NASH

     Or Oesophageal varices with high risk of bleeding :

     Size > 5 mm (stage 2 or 3) Or Size ≤ 5 mm and red spots Or Size ≤ 5 mm and Child-Pugh score C
  2. and/or the presence of a radiological sign of portal hypertension : Portosystemic shunts: rectal varices, splenorenal shunts, repermeabilization of the umbilical vein.
  3. and/or splenic elasticity > 50 kPa.
* Patients naive to treatment with cardioselective beta blockers
* Affiliated to french health insurance system

Exclusion Criteria:

* Absolute contraindications to beta blockers :

  * hypersensitivity to the active substance (carvedilol) or to any of the excipients listed in section 6.1 of the summary of product characteristics
  * patients with severe decompensated heart failure, with signs of fluid overload (oedema, ascites, pulmonary stasis rales), and/or requiring treatment with a positive inotrope or venous vasodilator
  * second and third-degree atrioventricular blocks (unless presence of a permanent pacemaker)
  * severe bradycardia (≤ 50 bpm)
  * cardiac sinus disease (including sino-auricular block)
  * severe hypotension (systolic pressure < 85 mm Hg)
  * cardiogenic shock
  * severe asthma, severe chronic obstructive pulmonary disease, history of severe bronchospasm
  * history of anaphylactic reaction
  * Raynaud's phenomenon
  * peripheral circulatory disorder: severe obliterative arterial disease of the lower limbs
  * association with cimetidine
  * association with class I antiarrhythmics except lidocaine
  * pulmonary arterial hypertension
* Presence of severe acute alcoholic hepatitis (Madrey score ≥ 32).
* Current hepatic encephalopathy ≥ Grade 2.
* Ongoing hepato-renal syndrome.
* Profuse clinical ascites (only if it interferes with the feasibility of echo-endoscopy).
* History of oesophageal varices rupture.
* Hepatocellular carcinoma active or in remission for less than six months.
* Active or resolved portal vein thrombosis for less than six months.
* History of digestive surgery that does not allow the porto-systemic gradient to be measured using echo-endoscopy (gastrectomy, by-pass, etc.).
* Patients taking antiaggregants (except acetylsalicylic acid) or anticoagulants for embologenic CA/FA.
* Severe stage 4 chronic renal insufficiency or stage 5 end-stage renal insufficiency (clearance < 30 mL/min).
* Pregnant or breast-feeding women, or those planning to become pregnant*.

  *A pregnancy test will be carried out for women of childbearing potential, and the investigator will ensure that effective contraception is in place while Carvedilol is being taken and for 5 half-lives after stopping it.
* Patients protected by law (under guardianship, curatorship or safeguard of justice) or deprived of their freedom.
* Patients currently taking part in another clinical research protocol.
* Patients who do not understand French language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a reduction of at least 10% in the porto-systemic gradient | One month after starting carvedilol.
  Hemodynamic response (binary efficacy criterion), defined as a reduction of at least 10% in the echo-endoscopic portosystemic gradient compared with the baseline value measured at inclusion.

SECONDARY OUTCOMES:
Side-effects of beta blockers | From enrollment to D90.
  Side effects of beta-blockers among the top ten reported in the literature, and percentage of patients discontinuing treatment due to side effects.
Number of participants with digestive hemorrhage | Within three months of starting Carvedilol.
  Digestive hemorrhage due to rupture of esophageal or gastric varices.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Abergel, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Lise Laclautre, Clermont-Ferrand
  - Chu Estaing Medecine Digestive Et Hepatobiliaire, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No